CLINICAL TRIAL: NCT00333411
Title: A 12 Week Double-blind, Randomised, Placebo-controlled, Modified Dose-escalation Trial to Investigate Safety, Efficacy, and Pharmacokinetics of BIRT 2584XX Tablets at Doses of 100, 300 and 500 mg Administered Once Daily in Patients With Moderate to Severe Psoriasis With a 12 Week Treatment Extension
Brief Title: Double-blind, Randomised, Placebo-controlled Trial Investigating BIRT 2584 XX in Patients With Moderate/Severe Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1206.5
Record Dates: First submitted 2006-06-02; First posted 2006-06-05 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-06

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

ARMS (4):
- BIRT 2584 XX high dose (Experimental)
  Interventions: Drug: BIRT 2584 XX
- BIRT 2584 XX medium dose (Experimental)
  Interventions: Drug: BIRT 2584 XX
- BIRT 2584 XX low dose (Experimental)
  Interventions: Drug: BIRT 2584 XX
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIRT 2584 XX
  Arms: BIRT 2584 XX high dose; BIRT 2584 XX low dose; BIRT 2584 XX medium dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this clinical study is to determine the effectiveness, pharmacokinetics and safety of several doses of BIRT 2584 XX (100mg, 300mg and 500mg) taken once daily in the treatment of moderate to severe plaque-type psoriasis. This new medicine will be compared to a so-called placebo medicine over 12 weeks with a 12 weeks treatment extension possible.

DETAILED DESCRIPTION:
The proposed study is a phase 2a/b international multicentre clinical trial. The general aim of this study is to investigate the safety and efficacy (clinical proof of concept) of three different doses (100 mg, 300 mg, or 500 mg) of BIRT 2584 XX tablets administered orally once daily compared to placebo tablets for the treatment of patients with moderate to severe plaque-type psoriasis patients who are candidates for systemic treatment or phototherapy. This study may also provide dose-finding information for future pivotal studies.

The response to treatment will be measured for all patients in the study after 12 weeks of treatment using the PASI as the primary endpoint, and also the sPGA. Both instruments evaluate the clinical severity of plaque-type psoriatic lesions. Training on PASI and sPGA assessment will be provided in order to decrease inter-observer variability. The sPGA is thus to be validated for future phase 3 trials.

After 12 weeks of treatment, only those patients with a response equivalent or better than PASI50 and with a satisfactory safety experience will enter a 12 week extension of the treatment period. The total time of exposure to study drug in this subgroup of patients will be 24 weeks. All other study patients will terminate treatment with study drug after 12 weeks.

In addition, the durability of remission/response, and the occurrence of any relapse or rebound during the treatment with study drug and after the end of treatment will be assessed in an 8 weeks follow-up period. The follow-up period is applicable to all study participants who have taken at least one dose of study drug. It initiates after the last dose of study medication has been taken, irrespective of the duration of the patients actual treatment period.

The trial will use a modified dose-escalation scheme. The randomisation to the 500 mg treatment arm will initiate only after a Data Safety Monitoring Board (DSMB) decision on the safety of the other treatment arms. An IVRS will be used for randomisation in this trial.

Ninety (90) patients are required per dose group. With four groups and an overall 1:1:1:1 randomisation scheme, a total of 360 eligible patients are planned to be randomised to treatment.

Study Hypothesis:

Psoriasis is a chronic inflammatory disease that leads to skin sores. These skin sores are dependent on the rate of growth of the skin which is driven by an underlying corresponding degree of local inflammation. The skin inflammation is caused by different cell types that move from the blood vessels into the skin. This cell movement is a result of interaction of different proteins. One of these proteins is called LFA-1 (Lymphocyte Function Associated Antigen 1). LFA-1 is then a promising target for psoriasis therapy. BIRT 2584 XX will block the passage of these inflammatory cells from the blood to the skin by blocking LFA-1, and thus indirectly block the inflammatory process. BIRT 2584 XX can also block the activation of local inflammatory cells, which altogether may reduce the signs and symptoms of psoriasis.

A dose-dependent effect of BIRT 2584 XX was observed on a set of markers in the blood that are believed to correlate with the severity of the inflammatory process leading to psoriasis.

Comparison(s):

In this clinical study, BIRT 2584 XX in a dose of 100 mg, 300 mg or 500 mg, or placebo will be given once daily. Patients will receive the same treatment throughout the study.

Patients will have a 1 in 4 chance (25%) of being allocated to placebo treatment. The placebo is identical in appearance compared to any one of the three dose groups with BIRT 2584 XX, but does not contain any active ingredient. The purpose of a comparison with placebo is to ensure a more reliable assessment of the therapeutic effect and of the side effects of BIRT 2584 XX.

ELIGIBILITY:
Inclusion_Criteria:

1. Age 18 to 75, males or females
2. Patients with stable moderate to severe plaque-type psoriasis involving ?10% body surface area, with minimum disease severity PASI ?10 and with static PGA of at least moderate (score of at least 3) at screening visit
3. Psoriasis disease duration of at least 6 months prior to screening
4. Patients must be candidates for systemic psoriasis treatment or phototherapy
5. Patient must give informed consent and sign an approved consent form prior to any study procedures, including wash out of prohibited medications (Patients participating in the PK sub-study will sign an additional consent form. Refusal to participate in the sub-study will not exclude from participation in the main trial)

Exclusion_Criteria:

1. Patients with primary guttatae, erythrodermic, or pustular psoriasis
2. Patients who have previously discontinued efalizumab treatment due to lack of efficacy
3. Patients using treatments that could interfere with the primary endpoint of the study (cf. protocol section 4.2.2.1)
4. Patients on treatment with warfarin, paracetamol (acetaminophen), some NSAIDs, some antidepressants, medications known to induce or inhibit CYP3A4, or any other concomitant medication where potential drug-drug interactions with BIRT 2584 XX could either result in decreased efficacy or an unacceptable benefit-risk assessment, and where replacement of that concomitant medication with a safe equivalent drug is not possible (cf. protocol section 4.2.2.2 and the Investigator Site File).
5. Patients with active liver disease or history of any significant liver disease.
6. Any clinically significant illness or unstable disease which according to investigator judgement may either put the patient at risk because of participation in the study or may influence the results of the study or the patients ability to participate.
7. Patient with serum creatinine and/or white blood cell count >1.5 x ULN at screening.

   (Repeat laboratory is allowed once between screening and randomisation prior to excluding the patient)
8. Patients with ALT, AST and/or total bilirubin > 1.5xULN at screening (Repeat laboratory is allowed once between screening and randomisation prior to excluding the patient)
9. Abnormal values of other laboratory parameters at screening that would define a clinically significant disease as described in # 6 above (Repeat laboratory is allowed once between screening and randomisation prior to excluding the patient)
10. Positive testing at screening, or history of HIV or hepatitis B or hepatitis C, or any serious infection (requiring hospitalisation or parenteral antibiotic therapy) in the past 3 months prior to screening
11. History of malignancy in the past 5 years or suspicion of active malignant disease except treated cutaneous squamous cell or basal cell carcinoma
12. Patients with the following findings at the screening visit that could interfere with cardiac repolarisation:

    * marked baseline prolongation of QT/QTc interval as measured on ECG (e.g. QTc interval >450ms);
    * history of additional risk factors for Torsade de pointe (e.g. heart failure, - hypokalemia, family history of long QT syndrome);
    * use of concomitant medications that prolong the QT/QTc interval
13. History of drug or alcohol abuse within the past two years
14. Pre-menopausal (last menstruation ≤ 1 year prior to screening) sexually active woman who:

    * is pregnant or nursing
    * is of child bearing potential and not practicing acceptable methods of birth control, or does not plan to continue practising an acceptable method throughout the study (acceptable methods of birth control include surgical sterilisation, intrauterine devices, double barrier, male partner sterilisation, but not hormonal contraceptives**) [A negative serum pregnancy test at screening (Visit 1) and a negative urine test prior to randomisation (Visit 2) are required]
15. Patient not willing to avoid excess sun exposure during the trial duration
16. Patients who have taken an investigational drug, within the last 4 weeks or 5 half lives (which ever is greater) prior to randomisation [Patients who have been treated with any investigational antibody or fusion protein within the past 12 weeks before randomisation are excluded]
17. Known allergy to BIRT 2584 XX or to the excipients used for tablet formulation
18. Body mass index > 34 kg/m2 at screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2006-06; Primary Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Achievement of > 75% reduction from baseline in Psoriasis Area and Severity Index (PASI) score (PASI75 ) at 12 weeks | 12 weeks

SECONDARY OUTCOMES:
Other PASI assessments, NPF Psoriasis Score Static Psoriasis Global Assessment (sPGA), Discontinuations of therapy due to lack of efficacy, Relapse and rebound, Dermatology Life Quality Index, Pain Visual Analog Scale for psoriatic arthritis | 12 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — BI France S.A.S.
Locations (47):
- Belgium (3):
  - Dermatologie Kliniek, Antwerp
  - Hôpital Erasme, Brussels
  - UZ Antwerpen, Edegem
- Canada (10):
  - Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - Eastern Canada Cutaneous Research Associates Ltd., Halifax, Nova Scotia
  - Boehringer Ingelheim Investigational Site, London, Ontario
  - Boehringer Ingelheim Investigational Site, Markham, Ontario
  - Boehringer Ingelheim Investigational Site, Waterloo, Ontario
  - Innovaderm Research Inc., Montreal, Quebec
  - Dr. Wayne Carey, Montreal, Quebec
  - Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - Boehringer Ingelheim Investigational Site, Sainte-Foy, Quebec
- Denmark (3):
  - Marselisborg Centret, Aarhus C
  - Amtssygehuset i Gentofte, Hellerup
  - Odense Universitetshospital, Odense C
- Päijät-Hämeen keskussairaala, Lahti, Finland
- France (6):
  - Hôpital Saint Jacques, Besançon
  - Hôpital Dupuytren, Limoges
  - Hôpital de L'Archet, Nice
  - Hôpital Saint Louis, Paris
  - CHU - Hôpital Nord, Saint-Priest-en-Jarez
  - Hôpital Nord, Saint-Priest-en-Jarez
- Germany (11):
  - Charite, Campus Virchow-Klinikum, Berlin
  - St. Josef-Hospital, Bochum
  - Universitätsklinikum an der TU Dresden, Dresden
  - Universitätsklinikum Erlangen, Erlangen
  - Universitäts-Hautklinik, Freiburg im Breisgau
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Otto-von-Guericke-Universität Magdeburg, Magdeburg
  - Boehringer Ingelheim Investigational Site, Mahlow
  - Johannes Gutenberg-Universität Mainz, Mainz
  - Universitätsklinikum Münster, Münster
  - Universitätsklinikum Ulm, Ulm
- Netherlands (2):
  - Academic Medical Centre, Amsterdam
  - University Medical Centre Nijmegen St. Radboud West, Nijmegen
- Spain (2):
  - Boehringer Ingelheim Investigational Site, Barcelona
  - Servicio de Dermatología, Madrid
- Karolinska Universitetssjukhuset Solna, Stockholm, Sweden
- United Kingdom (8):
  - Aberdeen Royal Infirmary, Department of Dermatology, Aberdeen
  - Cardiff University, Dermatology Department, Cardiff
  - Western Infirmary, Department of Dermatology, Glasgow
  - Royal Free Hospital, Dermatology Department,, London
  - Skin Therapy Research Unit, St John's Inst of Dermatolology, London
  - George Eliot Hospital, Dermatology Department, Nuneaton
  - Hope Hospital, The Dermatology Centre,, Salford
  - Royal South Hants Hospital, Dept of Dermatology, Southampton